CLINICAL TRIAL: NCT02321800
Title: A Multicenter, Double-blind, Randomized, Clinical Study to Assess the Efficacy and Safety of Intravenous S-649266 in Complicated Urinary Tract Infections With or Without Pyelonephritis or Acute Uncomplicated Pyelonephritis Caused by Gram-Negative Pathogens in Hospitalized Adults in Comparison With Intravenous Imipenem/Cilastatin
Brief Title: A Study of Efficacy and Safety of Intravenous Cefiderocol (S-649266) Versus Imipenem/Cilastatin in Complicated Urinary Tract Infections
Acronym: APEKS-cUTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1409R2121
Expanded Access: NCT03780140 (Approved for marketing)
Record Dates: First submitted 2014-11-11; First posted 2014-12-22 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Urinary Tract Infections
Keywords: S-649266; complicated urinary tract infection; cefiderocol; acute uncomplicated pyelonephritis; Gram-negative pathogens; imipenem/cilastatin
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cefiderocol; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefiderocol (Experimental): Participants received 2 g cefiderocol by intravenous injection once every 8 hours for 7 to 14 days.
  Interventions: Drug: Cefiderocol
- Imipenem/cilastatin (Active Comparator): Participants received 1 g each of imipenem/cilastatin by intravenous injection once every 8 hours for 7 to 14 days.
  Interventions: Drug: Imipenem/cilastatin

INTERVENTIONS:
Drug: Cefiderocol — 2000 mg intravenously every 8 hours for 7 to 14 days; dose adjustments for participants with reduced renal function (estimated CrCl ≤ 70 mL/minute) and/or body weight (< 70 kg) included every 6-hour dosing intervals and/or reduced doses.
  Other Names: FETROJA®; S-649266
  Arms: Cefiderocol
Drug: Imipenem/cilastatin — 1000 mg of each intravenously every 8 hours for 7 to 14 days; dose adjustments for participants with reduced renal function (estimated CrCl ≤ 70 mL/minute) and/or body weight (< 70 kg) included every 6-hour dosing intervals and/or reduced doses.
  Other Names: PRIMAXIN®
  Arms: Imipenem/cilastatin

SUMMARY:
The purpose of this study was to determine the efficacy and safety of intravenous cefiderocol (S-649266) in hospitalized adults with complicated urinary tract infections caused by Gram-negative pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male and female patients ≥ 18 years
* Clinical diagnosis of either complicated urinary tract infections (cUTI) with or without pyelonephritis or acute uncomplicated pyelonephritis
* cUTI diagnosed with a history of ≥ 1 of the following:

  * Indwelling urinary catheter or recent instrumentation of the urinary tract
  * Urinary retention (caused by benign prostatic hypertrophy)
  * Urinary retention of at least 100 mL or more of residual urine after voiding (neurogenic bladder)
  * Obstructive uropathy
  * Azotemia caused by intrinsic renal disease (blood urea nitrogen and creatinine values greater than normal laboratory values) OR Pyelonephritis and normal urinary tract anatomy, ie, acute uncomplicated pyelonephritis AND

At least 2 of the following signs or symptoms:

* Chills or rigors or warmth associated with fever (temperature greater than or equal to 38 degrees Celsius)
* Flank pain (pyelonephritis) or suprapubic/pelvic pain (cUTI)
* Nausea or vomiting
* Dysuria, urinary frequency, or urinary urgency
* Costo-vertebral angle tenderness on physical examination AND

All subjects had to have urinalysis evidence of pyuria demonstrated by 1 of the following:

* Dipstick analysis positive for leukocyte esterase
* ≥ 10 white blood cells (WBCs) per μL in unspun urine, or ≥ 10 WBCs per high power field in spun urine

  * Positive urine culture within 48 hours prior to randomization containing ≥10^5 colony forming unit (CFU)/mL of a Gram-negative uropathogen likely to be susceptible to imipenem (IPM)
  * Patients who were treated previously with an empiric antibiotic other than the study drugs but failed treatment, both clinically and microbiologically, were eligible for the study if they had an identified Gram-negative uropathogen that was not susceptible to the previously used empiric treatment and likely to be susceptible to IPM
  * Subjects receiving antibiotic prophylaxis for UTI who present with signs and symptoms consistent with an active new UTI

Exclusion Criteria:

* Urine culture identifies only a Gram-positive pathogen and/or a Gram-negative uropathogen resistant to IPM
* Urine culture at study entry isolates more than 2 uropathogens or patient has a confirmed fungal UTI
* Asymptomatic bacteriuria, the presence of >10^5 CFU/mL of a uropathogen and pyuria but without local or systemic symptoms
* Patient is receiving hemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

REFERENCES:
- [Result] Portsmouth S, van Veenhuyzen D, Echols R, Machida M, Ferreira JCA, Ariyasu M, Tenke P, Nagata TD. Cefiderocol versus imipenem-cilastatin for the treatment of complicated urinary tract infections caused by Gram-negative uropathogens: a phase 2, randomised, double-blind, non-inferiority trial. Lancet Infect Dis. 2018 Dec;18(12):1319-1328. doi: 10.1016/S1473-3099(18)30554-1. Epub 2018 Oct 25. PMID 30509675
- [Derived] Portsmouth S, Echols R, Toyoizumi K, Tillotson G, Nagata TD. Structured patient interview to assess clinical outcomes in complicated urinary tract infections in the APEKS-cUTI study: pilot investigation. Ther Adv Infect Dis. 2021 Nov 24;8:20499361211058257. doi: 10.1177/20499361211058257. eCollection 2021 Jan-Dec. PMID 34868583
- [Derived] Wenzler E, Butler D, Tan X, Katsube T, Wajima T. Pharmacokinetics, Pharmacodynamics, and Dose Optimization of Cefiderocol during Continuous Renal Replacement Therapy. Clin Pharmacokinet. 2022 Apr;61(4):539-552. doi: 10.1007/s40262-021-01086-y. Epub 2021 Nov 18. PMID 34792787
- [Derived] Naseer S, Weinstein EA, Rubin DB, Suvarna K, Wei X, Higgins K, Goodwin A, Jang SH, Iarikov D, Farley J, Nambiar S. US Food and Drug Administration (FDA): Benefit-Risk Considerations for Cefiderocol (Fetroja(R)). Clin Infect Dis. 2021 Jun 15;72(12):e1103-e1111. doi: 10.1093/cid/ciaa1799. PMID 33393598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 67 hospitals in 15 countries. Participants diagnosed with complicated urinary tract infections (cUTIs) with or without pyelonephritis or acute uncomplicated pyelonephritis were enrolled from February 5, 2015 to August 16, 2016.
Pre-assignment Details: Participants were randomly assigned (2:1) to receive either cefiderocol or imipenem-cilastatin. Randomization was stratified by clinical diagnosis (complicated urinary tract infection with or without pyelonephritis or with acute uncomplicated pyelonephritis) and region (North America, Europe, Russia, and Japan).
Period: Overall Study
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Started | 303 | 149
Received Study Drug | 300 | 148
Completed | 283 | 138
Not Completed | 20 | 11
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 10 | 4
Not completed — Adverse Event | 2 | 3
Not completed — Other, Miscellaneous | 3 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat population includes all randomly assigned participants who received at least one dose of study drug and had qualifying Gram-negative uropathogen (≥1 × 10⁵ colony forming unit (CFU)/mL)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefiderocol | Imipenem/Cilastatin | Total
Number analyzed (Participants) | 252 | 119 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (16.10) | 61.3 (18.48) | 62.0 (16.88)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 113 | 54 | 167
  >= 65 years | 139 | 65 | 204
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 71 | 204
  Male | 119 | 48 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 247 | 118 | 365
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 241 | 115 | 356
  Black or African American | 1 | 0 | 1
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
Creatinine Clearance Renal Grading Group [Count of Participants; unit: Participants] — Creatinine clearance was calculated using the Cockcroft-Gault formula ([140 - age in years] × [weight in kg])/(72 × serum creatinine in mg/dL [multiplied by 0·85 for women]) using data from the central laboratory. Population: Participants with available data
  Participants
    number analyzed (Participants) | 250 | 119 | 369
    > 80 mL/min (Normal) | 124 | 51 | 175
    > 50 - 80 mL/min (Mild) | 78 | 41 | 119
    30 - 50 mL/min (Moderate) | 41 | 23 | 64
    < 30 mL/min (Severe) | 7 | 4 | 11
Clinical Diagnosis at Baseline [Count of Participants; unit: Participants]
  cUTI with pyelonephritis | 65 | 29 | 94
  cUTI without pyelonephritis | 122 | 55 | 177
  Acute Uncomplicated Pyelonephritis | 65 | 35 | 100
Number of Gram-negative Uropathogens > 10⁵ CFU/mL Isolated at Baseline [Count of Participants; unit: Participants]
  1 uropathogen | 241 | 115 | 356
  2 uropathogens | 11 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Test of Cure
Description: The primary efficacy endpoint was the composite outcome of clinical response and microbiological response at the test of cure assessment, defined as 7 days (±2 days) after the end of antibiotic treatment.
  Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with response defined as resolution or improvement of complicated urinary tract infection symptoms present at study entry and the absence of new symptoms.
  Microbiological outcome was based on quantitative microbiological urine cultures, with eradication defined as the bacterial pathogen found at study entry at > 1 × 10⁵ CFU/mL reduced to 1 × 10⁴ CFU/mL or less.
Time Frame: Test of cure (TOC; 7 days after end of treatment [EOT], equivalent to Study Day 14 to 21)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 72.6 | 54.6
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; Adjusted estimates of the difference between the two treatment groups are based on a stratified analysis using Cochran-Mantel-Haenszel weights, with clinical diagnosis (complicated urinary tract infection with or without pyelonephritis vs acute uncomplicated pyelonephritis) as the stratification factor; Test type: Non-Inferiority — The margin of noninferiority was 20%. Noninferiority was concluded if the lower bound of a 2-sided 95% CI for the difference in response rates between the 2 treatment groups was greater than -20%. If the noninferiority inference based on the 20% margin was concluded successfully, noninferiority inference based on the 15% margin was performed; Treatment Difference = 18.58, 95% CI 2-sided [8.23 to 28.92]

2. Secondary Outcome: Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Early Assessment
Description: A composite outcome of clinical response and microbiological response at the early assessment, defined as Day 4 of antibiotic treatment.
  Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with response defined as resolution or improvement of complicated urinary tract infection symptoms present at study entry and the absence of new symptoms.
  Microbiological outcome was based on quantitative microbiological urine cultures, with eradication defined as the bacterial pathogen found at study entry at > 1 × 10⁵ CFU/mL reduced to 1 × 10⁴ CFU/mL or less.
Time Frame: Early assessment (EA; Day 4)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 88.1 | 87.4
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 0.66, 95% CI 2-sided [-6.48 to 7.79]

3. Secondary Outcome: Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at End of Treatment
Description: A composite outcome of clinical response and microbiological response at the end of treatment, defined as the end of the last infusion of antibiotic treatment.
  Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with response defined as resolution or improvement of complicated urinary tract infection symptoms present at study entry and the absence of new symptoms.
  Microbiological outcome was based on quantitative microbiological urine cultures, with eradication defined as the bacterial pathogen found at study entry at > 1 × 10⁵ CFU/mL reduced to 1 × 10⁴ CFU/mL or less.
Time Frame: End of treatment (EOT; Day 7 to 14)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 96.4 | 95.8
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 0.72, 95% CI 2-sided [-3.48 to 4.92]

4. Secondary Outcome: Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Follow-up
Description: A composite response of clinical response and microbiological response at the follow-up assessment, defined as 14 days after the end of treatment.
  Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with sustained response defined as all pre-therapy signs and symptoms of cUTI show no evidence of recurrence after administration of the last dose of study drug.
  Microbiological outcome was based on quantitative microbiological urine cultures, with sustained eradication defined as a urine culture obtained after documented eradication at the TOC, up to and including the FUP, showed that the bacterial uropathogen(s) identified at baseline at ≥ 10⁵ CFU/mL remained < 10⁴ CFU/mL.
Time Frame: Follow-up (FUP; 14 days after end of treatment, Day 21 to 28)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 54.4 | 39.5
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; Test type: Other; Treatment Difference = 15.31, 95% CI 2-sided [4.69 to 25.92]

5. Secondary Outcome: Percentage of Participants With Microbiological Eradication at Test of Cure
Description: Microbiological outcome was based on quantitative microbiological urine cultures, with eradication defined as all bacterial uropathogens found at study entry at > 1 × 10⁵ CFU/mL reduced to 1 × 10⁴ CFU/mL or less.
Time Frame: Test of cure (7 days after end of treatment, Day 14 to 21)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 73.0 | 56.3
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 17.25, 95% CI 2-sided [6.92 to 27.58]

6. Secondary Outcome: Percentage of Participants With Microbiological Eradication at Early Assessment
Description: as for outcome 5
Time Frame: Early assessment, Day 4
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 92.1 | 90.8
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 1.28, 95% CI 2-sided [-4.83 to 7.39]

7. Secondary Outcome: Percentage of Participants With Microbiological Eradication at End of Treatment
Description: as for outcome 5
Time Frame: End of treatment, Day 7 to 14
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 96.8 | 95.8
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 1.10, 95% CI 2-sided [-3.04 to 5.25]

8. Secondary Outcome: Percentage of Participants With Microbiological Eradication at Follow-up
Description: Microbiological outcome was based on quantitative microbiological urine cultures, with sustained eradication defined as a urine culture obtained after documented eradication at the TOC, up to and including the FUP, where the bacterial uropathogen(s) identified at baseline at ≥ 10⁵ CFU/mL remained < 10⁴ CFU/mL.
Time Frame: Follow-up, 14 days after end of treatment, Day 21 to 28
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 57.1 | 43.7
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 13.92, 95% CI 2-sided [3.21 to 24.63]

9. Secondary Outcome: Percentage of Participants With Microbiological Eradication at Test of Cure Per Uropathogen
Description: Microbiological outcome was based on quantitative microbiological urine cultures, with eradication defined as the bacterial pathogen found at study entry at > 1 × 10⁵ CFU/mL reduced to 1 × 10⁴ CFU/mL or less.
  Results are reported for the 4 most frequent uropathogens, Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, and Proteus mirabilis.
Time Frame: Test of cure; 7 days after end of treatment, Day 14 to 21
Population: Modified intent-to-treat population with the relevant pathogen at Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 231 | 110
percentage of participants
  Escherichia coli: number analyzed (Participants) | 152 | 79
  Escherichia coli | 75.0 | 58.2
  Klebsiella pneumoniae: number analyzed (Participants) | 48 | 25
  Klebsiella pneumoniae | 75.0 | 52.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 18 | 5
  Pseudomonas aeruginosa | 44.4 | 60.0
  Proteus mirabilis: number analyzed (Participants) | 17 | 2
  Proteus mirabilis | 76.5 | 50.0

10. Secondary Outcome: Percentage of Participants With Microbiological Eradication at Early Assessment Per Uropathogen
Description: as for outcome 9
Time Frame: Early assessment, Day 4
Population: Intent-to-treat population with the relevant pathogen at Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 231 | 110
percentage of participants
  Escherichia coli: number analyzed (Participants) | 152 | 79
  Escherichia coli | 92.8 | 94.9
  Klebsiella pneumoniae: number analyzed (Participants) | 48 | 25
  Klebsiella pneumoniae | 89.6 | 88.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 18 | 5
  Pseudomonas aeruginosa | 94.4 | 80.0
  Proteus mirabilis: number analyzed (Participants) | 17 | 2
  Proteus mirabilis | 88.2 | 100.0

11. Secondary Outcome: Percentage of Participants With Microbiological Eradication at End of Treatment Per Uropathogen
Description: as for outcome 9
Time Frame: End of treatment, Day 7 to 14
Population: Modified intent-to-treat population with the relevant pathogen at Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 231 | 110
percentage of participants
  Escherichia coli: number analyzed (Participants) | 152 | 79
  Escherichia coli | 98.7 | 97.5
  Klebsiella pneumoniae: number analyzed (Participants) | 48 | 25
  Klebsiella pneumoniae | 97.9 | 92.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 18 | 5
  Pseudomonas aeruginosa | 88.9 | 100.0
  Proteus mirabilis: number analyzed (Participants) | 17 | 2
  Proteus mirabilis | 94.1 | 100.0

12. Secondary Outcome: Percentage of Participants With Microbiological Eradication at Follow-up Per Uropathogen
Description: Microbiological outcome was based on quantitative microbiological urine cultures, with sustained eradication defined as a urine culture obtained after documented eradication at the TOC, up to and including the FUP, where the bacterial uropathogen identified at baseline at ≥ 10⁵ CFU/mL remained < 10⁴ CFU/mL.
  Results are reported for the 4 most frequent uropathogens, Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, and Proteus mirabilis.
Time Frame: Follow-up, 14 days after the end of treatment, Day 21 to 28
Population: Modified intent-to-treat population with the relevant pathogen at Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 231 | 110
percentage of participants
  Escherichia coli: number analyzed (Participants) | 152 | 79
  Escherichia coli | 59.9 | 41.8
  Klebsiella pneumoniae: number analyzed (Participants) | 48 | 25
  Klebsiella pneumoniae | 58.3 | 52.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 18 | 5
  Pseudomonas aeruginosa | 27.8 | 20.0
  Proteus mirabilis: number analyzed (Participants) | 17 | 2
  Proteus mirabilis | 64.7 | 0

13. Secondary Outcome: Percentage of Participants With Clinical Response at Test of Cure
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with response defined as resolution or improvement of complicated urinary tract infection symptoms present at study entry and the absence of new symptoms.
Time Frame: Test of cure, 7 days after end of treatment, Day 14 to 21
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 89.7 | 87.4
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 2.39, 95% CI 2-sided [-4.66 to 9.44]

14. Secondary Outcome: Percentage of Participants With Clinical Response at Early Assessment
Description: as for outcome 13
Time Frame: Early assessment, Day 4
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 90.5 | 90.8
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = -0.26, 95% CI 2-sided [-6.57 to 6.05]

15. Secondary Outcome: Percentage of Participants With Clinical Response at End of Treatment
Description: as for outcome 13
Time Frame: End of treatment, Day 7 to 14
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 98.0 | 99.2
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = -1.07, 95% CI 2-sided [-3.42 to 1.29]

16. Secondary Outcome: Percentage of Participants With Clinical Response at Follow-up
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with sustained response defined as all pre-therapy signs and symptoms of cUTI showing no evidence of recurrence after administration of the last dose of study drug.
Time Frame: Follow-up, 14 days after end of treatment, Day 21 to 28
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 252 | 119
percentage of participants | 81.3 | 72.3
Statistical Analysis 1: Comparison: Cefiderocol vs Imipenem/Cilastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Treatment Difference = 9.02, 95% CI 2-sided [-0.37 to 18.41]

17. Secondary Outcome: Percentage of Participants With Clinical Response at Test of Cure Per Uropathogen
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with response defined as resolution or improvement of complicated urinary tract infection symptoms present at study entry and the absence of new symptoms. Results are reported for the 4 most frequent uropathogens, Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, and Proteus mirabilis.
Time Frame: Test of cure, 7 days after end of treatment, Day 14 to 21
Population: Modified intent-to-treat population with the relevant pathogen at Baseline and available clinical outcome data
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 220 | 107
percentage of participants
  Escherichia coli: number analyzed (Participants) | 146 | 77
  Escherichia coli | 89.7 | 88.3
  Klebsiella pneumoniae: number analyzed (Participants) | 46 | 25
  Klebsiella pneumoniae | 89.1 | 84.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 15 | 4
  Pseudomonas aeruginosa | 73.3 | 75.0
  Proteus mirabilis: number analyzed (Participants) | 13 | 1
  Proteus mirabilis | 100.0 | 100.0

18. Secondary Outcome: Percentage of Participants With Clinical Response at Early Assessment Per Uropathogen
Description: as for outcome 17
Time Frame: Early assessment, Day 4
Population: Modified intent-to-treat population with the relevant pathogen at Baseline and with available clinical outcome data
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 220 | 107
percentage of participants
  Escherichia coli: number analyzed (Participants) | 146 | 77
  Escherichia coli | 91.8 | 96.1
  Klebsiella pneumoniae: number analyzed (Participants) | 46 | 25
  Klebsiella pneumoniae | 82.6 | 88.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 15 | 4
  Pseudomonas aeruginosa | 93.3 | 75.0
  Proteus mirabilis: number analyzed (Participants) | 13 | 1
  Proteus mirabilis | 84.6 | 100.0

19. Secondary Outcome: Percentage of Participants With Clinical Response at End of Treatment Per Uropathogen
Description: as for outcome 17
Time Frame: End of treatment, Day 7 to 14
Population: Modified intent-to-treat population with the relevant pathogen at Baseline and with available clinical outcome data
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 220 | 107
percentage of participants
  Escherichia coli: number analyzed (Participants) | 146 | 77
  Escherichia coli | 97.9 | 98.7
  Klebsiella pneumoniae: number analyzed (Participants) | 46 | 25
  Klebsiella pneumoniae | 100.0 | 100.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 15 | 4
  Pseudomonas aeruginosa | 93.3 | 100.0
  Proteus mirabilis: number analyzed (Participants) | 13 | 1
  Proteus mirabilis | 100.0 | 100.0

20. Secondary Outcome: Percentage of Participants With Clinical Response at Follow-up Per Uropathogen
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms, with sustained response defined as all pre-therapy signs and symptoms of cUTI show no evidence of recurrence after administration of the last dose of study drug. Results are reported for the 4 most frequent uropathogens, Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, and Proteus mirabilis.
Time Frame: Follow-up, 14 days after the end of treatment, Day 21 to 28
Population: Modified intent-to-treat population with the relevant pathogen at Baseline and with available clinical outcome data
Measure: Number; unit: percentage of participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 220 | 107
percentage of participants
  Escherichia coli: number analyzed (Participants) | 146 | 77
  Escherichia coli | 82.9 | 72.7
  Klebsiella pneumoniae: number analyzed (Participants) | 46 | 25
  Klebsiella pneumoniae | 82.6 | 68.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 15 | 4
  Pseudomonas aeruginosa | 53.3 | 75.0
  Proteus mirabilis: number analyzed (Participants) | 13 | 1
  Proteus mirabilis | 84.6 | 100.0

21. Secondary Outcome: Plasma Concentration of Cefiderocol
Time Frame: On Day 3 of dosing prior to infusion, end of infusion, and at 1 hour post infusion
Population: The pharmacokinetic (PK) concentration population included all participants who underwent plasma or urine PK sampling and had at least 1 evaluable PK assay result for cefiderocol
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cefiderocol
Number analyzed (Participants) | 293
µg/mL
  Pre-infusion: number analyzed (Participants) | 232
  Pre-infusion | 18.0 (18.3)
  End of infusion: number analyzed (Participants) | 190
  End of infusion | 141 (220)
  1 hour after end of infusion: number analyzed (Participants) | 214
  1 hour after end of infusion | 70.2 (30.4)

22. Secondary Outcome: Urine Concentration of Cefiderocol
Time Frame: Day 3, 2 hours and 6 hours after end of infusion
Population: Pharmacokinetic concentration population with available urine concentration data
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cefiderocol
Number analyzed (Participants) | 8
µg/mL
  2 hours after end of infusion | 2710 (1520)
  6 hours after end of infusion | 1520 (1370)

23. Secondary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event was defined by regulation as any adverse event (AE) occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening condition
  * Hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Other medically important condition.
  The relationship of an event to the study drug was determined by the investigator based on whether the AE could be reasonably explained as being caused by the study drug.
Time Frame: From first dose of study drug until 28 days after end of treatment; Day 35 to 42
Population: The safety population included all randomized participants who received at least 1 dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cefiderocol | Imipenem/Cilastatin
Number analyzed (Participants) | 300 | 148
Participants
  All adverse events | 122 | 76
  Drug-related adverse events | 27 | 17
  Deaths | 1 | 0
  Serious adverse events | 14 | 12
  Drug-related serious adverse events | 1 | 1
  Discontinuation of study drug due to AE | 5 | 3
  Discontinuation due to drug-related AE | 3 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 28 days after end of treatment; Day 35 to 42
Arm/Group | S-649266 | Imipenem/Cilastatin
All-Cause Mortality (participants affected / at risk) | 1/300 | 0/148
Serious Adverse Events (participants affected / at risk) | 14/300 | 12/148
Other Adverse Events (participants affected / at risk) | 60/300 | 48/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S-649266 (N=300) | Imipenem/Cilastatin (N=148)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Congenital ureteric anomaly (Congenital, familial and genetic disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Ascariasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Obstructive nephropathy (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urethrotomy (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S-649266 (N=300) | Imipenem/Cilastatin (N=148)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 12 | 8
Nausea (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 6 | 2
Infusion site erythema (General disorders) | 3 | 3
Infusion site pain (General disorders) | 9 | 5
Clostridium difficile colitis (Infections and infestations) | 0 | 3
Vaginal infection (Infections and infestations) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 4
Headache (Nervous system disorders) | 7 | 8
Insomnia (Psychiatric disorders) | 4 | 3
Renal cyst (Renal and urinary disorders) | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Hypertension (Vascular disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.